CLINICAL TRIAL: NCT02477397
Title: Effectiveness of Single Inhaler Maintenance and Reliever Therapy With Spiromax® Budesonide/Formoterol (SMART) Versus Fixed Dose Treatment With Diskus® Fluticasone/Salmeterol in Patients With a Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Symptom-driven Maintenance and Reliever Treatment to Prevent Exacerbations in COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, Dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART2014
Record Dates: First submitted 2015-05-28; First posted 2015-06-22 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: COPD
Keywords: Spiromax; Budesonide/formoterol; COPD; exacerbations; SMART
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spiromax Budesonide/formoterol (Experimental): 1. In Group A, Patients will be treated with Spiromax® budesonide/formoterol 160/4.5 μg two inhalations twice daily + Spiromax® budesonide/formoterol 160/4.5 μg as needed with a maximum of 8 additional inhalations daily.
  Interventions: Drug: Spiromax Budesonide/formoterol
- Diskus Fluticasone/salmeterol (Active Comparator): 2. In group B, Patients will be treated with Diskus® fluticasone/salmeterol 500/50 μg one inhalation twice daily + salbutamol 100 μg as needed with a maximum of 8 inhalations daily.
  Interventions: Drug: Diskus Fluticasone/salmeterol

INTERVENTIONS:
Drug: Spiromax Budesonide/formoterol — 1. In Group A, Patients will be treated with Spiromax® budesonide/formoterol 160/4.5 μg two inhalations twice daily + Spiromax® budesonide/formoterol 160/4.5 μg as needed with a maximum of 8 additional inhalations daily.
  Other Names: Spiromax® budesonide/formoterol
  Arms: Spiromax Budesonide/formoterol
Drug: Diskus Fluticasone/salmeterol — 2. In group B, Patients will be treated with Diskus® fluticasone/salmeterol 500/50 μg one inhalation twice daily + salbutamol 100 μg as needed with a maximum of 8 inhalations daily.
  Other Names: Diskus® Fluticasone/salmeterol
  Arms: Diskus Fluticasone/salmeterol

SUMMARY:
Study to investigate the effects of symptom-driven maintenance and reliever therapy in COPD.

DETAILED DESCRIPTION:
Rationale: Chronic obstructive pulmonary disease (COPD) is a leading cause of death worldwide and its morbidity and mortality are still rising. A symptom-driven maintenance and reliever therapy (SMART) with budesonide/formoterol is a frequently used treatment strategy in asthma. Several studies have shown that the SMART approach effectively reduces the number of asthma exacerbations when compared to a fixed maintenance dose of, e.g. fluticasone/salmeterol. In addition, larger improvements in lung function and symptoms have been observed in asthma patients with the SMART approach. Thus far, no studies have investigated the efficacy of the SMART approach in patients with COPD. The investigators hypothesize that SMART treatment with budesonide/formoterol will be more effective than fluticasone/salmeterol fixed dose treatment in COPD.

Objective: This research proposal aims to investigate the efficacy of the SMART approach with budesonide/fomoterol versus fixed dose treatment with fluticasone/salmeterol in patients with COPD.

Study design: This will be a randomized, parallel 2-arm, open-label, multi-centre study.

Study population: A total of 260 COPD patients will be included with a smoking history of >10 pack years, an FEV1 <80% predicted either or not using inhaled corticosteroids and having had at least one COPD exacerbation during the 2 years prior to inclusion.

Intervention: COPD patients will be randomized to one of the following two treatment groups:

A: One year Spiromax® budesonide/formoterol 160/4.5 μg two inhalations twice daily + Spiromax® budesonide/formoterol 160/4.5 μg as needed with a maximum of 8 inhalations daily.

B: One year Diskus® fluticasone/salmeterol 500/50 μg one inhalation twice daily + salbutamol 100 μg as needed with a maximum of 8 inhalations daily.

Main study endpoints/objectives: The primary endpoint is the reduction in number of COPD exacerbations requiring treatment with oral prednisolone).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study has no specific benefits for the participating patients. The study also has no major risks. Minor risks for participants in this study are:

* Nasal epithelium collection may cause a temporary nose bleed.
* Blood collection may cause bruising.
* All drugs may cause side effects. The combination treatments with an inhaled corticosteroid and long-acting β2-agonist: budesonide/formoterol and fluticasone/salmeterol are medicinal products that have been on the market for many years in many countries and they are often prescribed both in asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years
* Smoking history of > 10 pack years
* COPD patients with an FEV1 < 80% predicted either or not using inhaled corticosteroids.
* At least one COPD exacerbation for which oral prednisolone had to be prescribed during 2 years prior to inclusion in the study

Exclusion Criteria:

* History of asthma.
* Exacerbation or respiratory tract infection during the last 4 weeks prior to randomization.
* Females of childbearing potential without an efficient contraception unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL or the use of one or more of the following acceptable methods of contraception:

  1. Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy).
  2. Hormonal contraception (implantable, patch, oral, injectable).
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository.
  4. Continuous abstinence.
* Periodic abstinence (e.g. calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception should be maintained throughout the study and for 30 days after study drug discontinuation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with increase in symptoms of dyspnea, cough, sputum production | 1 year

SECONDARY OUTCOMES:
Lung function FEV1 | 1 year

OTHER OUTCOMES:
Cell differential counts in blood | 1 year
  Inflammation
Symptoms Questionnaire (CCQ) | 1 year
Gene expression | 1 year
  nasal gene expression signature

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Wisselink HJ, Pelgrim GJ, Rook M, Dudurych I, van den Berge M, de Bock GH, Vliegenthart R. Improved precision of noise estimation in CT with a volume-based approach. Eur Radiol Exp. 2021 Sep 10;5(1):39. doi: 10.1186/s41747-021-00237-x. PMID 34505172